CLINICAL TRIAL: NCT00127062
Title: Health Effects of Diesel Exhaust in Asthmatic Patients: A Real-world Study in a London Street
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Health Effects Institute (Other)
Responsible Party: Principal Investigator, Fan Chung, Professor, Imperial College London
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 03-194
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Exposure to Oxford Street; Exposure to Hyde Park
MeSH Terms: conditions — Asthma | interventions — hemoglobin M Akita

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma (Experimental): Asthma patients ranging from mild to severe
  Interventions: Other: Oxford street; Other: Hyde park
- Healthy Non-Smokers (Other)
  Interventions: Other: Oxford street; Other: Hyde park

INTERVENTIONS:
Other: Oxford street — 2 h walk around Oxford street
Other: Hyde park — 2 h walk around Hyde park

SUMMARY:
Acute exposure to diesel exhaust under normal city conditions leads to a worsening of symptoms of asthma, with reduction in lung function in asthmatic nonsmoking adults, dependent on the exposure dose and on the background severity of asthma.

The worsening asthma is accompanied by increased oxidative stress and inflammation in the lungs.

DETAILED DESCRIPTION:
The investigators will recruit 60 nonsmoking asthmatics of mild and of moderate severity. They will be exposed to Oxford St. or to Hyde Park for 2 hours each, at a walking pace. Real time exposure to PM2.5, carbon monoxide and nitrogen dioxide will be made each time. Health outcome measurements will be made before and after exposure to each street. Statistical analyses will be made to examine the effect of diesel exposure on changes in health outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be selected according to the current severity of their asthma; thirty from Steps 1 and 2 and thirty from Step 3 of the World Health Organization (WHO) Global Initiative for Asthma (GINA) asthma guidelines. These will include mild and moderate asthmatic states. Depending on baseline FEV1, subjects will undergo either a methacholine bronchial hyperresponsiveness assessment or airways reversibility testing. Subjects with normal FEV1 (>80% predicted) or normal FEV1/FVC ratio will undergo methacholine challenge. Subjects with FEV1 <80% predicted will undergo airways reversibility testing. Subjects must have either a PC20 of less than 8mg/ml methacholine, or improvement in FEV1 of 12% or more, following inhalation of short acting β-agonist (salbutamol 200μg from metered dose inhaler [MDI]). Skin prick testing will be conducted for common allergens (house dust mite, grass pollen, aspergillus fumigatus and cat hair). The results will only be for descriptive purposes, not as subject inclusion/exclusion criteria. Subjects may be atopic or non-atopic (according to history and allergy testing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2003-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cullinan, MD, Principal Investigator — Imperial College London; Fan Chung, MD, Study Director — Imperial College London; Mark Nieuwenhuijsen, PhD, Principal Investigator — Imperial College London; Jim Zhang, PhD, Principal Investigator — Rutgers U & UMDNJ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang JJ, McCreanor JE, Cullinan P, Chung KF, Ohman-Strickland P, Han IK, Jarup L, Nieuwenhuijsen MJ. Health effects of real-world exposure to diesel exhaust in persons with asthma. Res Rep Health Eff Inst. 2009 Feb;(138):5-109; discussion 111-23. PMID 19449765

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy volunteers were not recruited. Only asthma patients.
Groups:
- Mild Asthma: Asthma patients with mild asthma
- Moderate Asthma: Asthma patients with moderate asthma
Period: First intervention_Oxford Street
Arm/Group | Mild Asthma | Moderate Asthma
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0
Period: Second intervention_Hyde Park
Arm/Group | Mild Asthma | Moderate Asthma
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Asthma | Moderate Asthma | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Full Range); unit: years] | 31 [20 to 49] | 34 [19 to 55] | 32 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 17 | 14 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Spirometry, Percentage Change in FEV1 From Baseline
Time Frame: baseline, 24 hours after
Measure: Mean (95% Confidence Interval); unit: percentage change in FEV1 from baseline
Groups:
- Mild Asthma Hyde Park: Mild asthma patients walking on Hyde park
- Mild Asthma Oxford Street: Mild asthma patients walking on Oxford Street
- Moderate Asthma Hyde Park: Moderate asthma patients walking on Hyde park
- Moderate Asthma Oxford Street: Moderate asthma patients walking on Oxford Street
Arm/Group | Mild Asthma Hyde Park | Mild Asthma Oxford Street | Moderate Asthma Hyde Park | Moderate Asthma Oxford Street
Number analyzed (Participants) | 31 | 31 | 29 | 29
percentage change in FEV1 from baseline | -1.0 [-3.0 to 0.6] | -4.8 [-6.8 to -2.8] | -2.2 [-4.0 to -1.0] | -7.4 [-9.5 to -5.5]
Statistical Analysis 1: Comparison: Moderate Asthma Hyde Park vs Moderate Asthma Oxford Street; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Mild Asthma Hyde Park vs Mild Asthma Oxford Street; Test type: Superiority; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 hours
Groups:
- Mild asthma_Oxford Street: Asthma patients with mild asthma walked at Oxford street
- Mild asthma_Hyde Park: Asthma patients with mild asthma walked at Hyde park
- Moderate asthma_Oxford Street: Asthma patients with moderate asthma walked at Oxford street
- Moderate asthma_Hyde Park: Asthma patients with moderate asthma walked at Hyde park
Arm/Group | Mild asthma_Oxford Street | Mild asthma_Hyde Park | Moderate asthma_Oxford Street | Moderate asthma_Hyde Park
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes